CLINICAL TRIAL: NCT03520517
Title: Open-Label Study to Evaluate Safety, Tolerability and Pharmacokinetics of Multiple Doses of BHV-0223 in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Open-label Study to Evaluate Safety, Tolerability and PK of BHV-0223 in ALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV0223-103
Record Dates: First submitted 2018-04-17; First posted 2018-05-09 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-02

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS; Lou Gehrig Disease; Lou Gehrig's Disease; Lou-Gehrigs Disease; Motor Neuron Disease, Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Biohaven; Motor Neuron Disease, Amyotrophic Lateral Sclerosis; Lou Gehrig's Disease; Lou-Gehrigs Disease; Lou Gehrig Disease; Riluzole; Rilutek®; Neuroprotective Agents; Administration, Sublingual; Administration, Oral; Biological Availability
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BHV-0223 (Experimental): riluzole 40 mg sublingual tablet
  Interventions: Drug: BHV-0223

INTERVENTIONS:
Drug: BHV-0223 — BHV-0223, 40 mg BID

SUMMARY:
Phase 1, open-label study of BHV-0223 in ALS.

DETAILED DESCRIPTION:
This is a phase 1, open-label, single arm study to evaluate the safety, tolerability and pharmacokinetics of multiple doses of BHV-0223 in subjects with ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with diagnosed ALS by the revised El Escorial diagnostic criteria, including laboratory supported probable, probable, or definite ALS;
2. Subjects who have never taken riluzole tablets, OR Subjects who previously took riluzole tablets but discontinued at least 1 month prior to the screening visit. Subjects must not have had ALT or AST > 5 x ULN while taking riluzole tablets, or any other clinically significant tolerability issues (e.g., hypersensitivity reactions) in the judgement of the investigator;
3. Subjects determined by the investigator to be medically stable;
4. Subjects determined by the investigator to be willing and physically able to complete the study as designed, with or without caregiver assistance.

Exclusion Criteria:

1. Target Disease Exceptions
2. Medical History Exceptions

   1. Subject is known to have a current diagnosis of acute or chronic viral hepatitis;
   2. Subject is known to have any other acute or chronic liver disease that is clinically significant in the investigator's judgment;
   3. Subject has a history of a clinically significant medical condition that would interfere with the subject's ability to comply with study instructions, would place the subject at increased risk, or might confound the interpretation of the study results in the investigator's judgment;
   4. Any other sound medical, psychiatric and/or social reason in the investigator's judgment;
3. Physical and Laboratory Test Findings

   1. Positive urine pregnancy test in WOCBP at screening;
   2. Subject has evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, or other determinations beyond what is consistent with the target population, in the investigator's judgment;
   3. Subject has liver function testing abnormalities (ALT, AST , or total bilirubin) that are > 1 x ULN;
4. Other Exclusions a. Subjects who are unable to be compliant with the visit schedule or protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) | Through Week 8 (Day 57)
  Incidence of treatment emergent adverse events (safety and tolerability) as measured through laboratory tests and physical exam findings.

SECONDARY OUTCOMES:
BHV-0223 Concentrations in Blood at Days 1, 29 and 57 | Through Week 8 (Day 57)
  BHV-0223 concentrations at days 1, 29 and 57 through blood collections at days 1, 29 and 57.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Holy Cross Neuroscience Research Institute, Fort Lauderdale, Florida
  - Somnos/Neurology Associates Clinical Research, Lincoln, Nebraska
  - Neurosciences Institute, Neurology - Charlotte, Charlotte, North Carolina
  - Wesley Neurology Clinic, Cordova, Tennessee
  - Texas Neurology, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No